CLINICAL TRIAL: NCT04708821
Title: DEXTENZA Versus Topical Steroid or Antihistamine Therapy for Treatment of Allergic Conjunctivitis
Brief Title: DEXTENZA Therapy for Treatment of Allergic Conjunctivitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinical Research Center of Florida (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Dex-AC Study
Record Dates: First submitted 2020-12-15; First posted 2021-01-14 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Bilateral Conjunctivitis (Disorder)
MeSH Terms: interventions — Calcium Dobesilate; Loteprednol Etabonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- DEXTENZA (Experimental): DEXTENZA (dexamethasone ophthalmic insert) 0.4 mg, for intracanalicular use
  Interventions: Drug: Dexamethasone ophthalmic insert 0.4Mg
- Antihistamine (Active Comparator): PAZEO (olopatadine hydrochloride ophthalmic solution) 0.7% for topical ophthalmic administration.
  Interventions: Drug: olopatadine hydrochloride ophthalmic solution 0.7%
- Topical Steroid (Active Comparator): ALREX® (loteprednol etabonate ophthalmic suspension) contains a sterile, topical anti-inflammatory corticosteroid for ophthalmic use.
  Interventions: Drug: 0.2% loteprednol etabonate ophthalmic suspension

INTERVENTIONS:
Drug: Dexamethasone ophthalmic insert 0.4Mg — Dextenza 0.4Mg Ophthalmic Insert
  Other Names: Dextenza
  Arms: DEXTENZA
Drug: 0.2% loteprednol etabonate ophthalmic suspension — 0.2% loteprednol etabonate ophthalmic suspension
  Other Names: ALREX
  Arms: Topical Steroid
Drug: olopatadine hydrochloride ophthalmic solution 0.7% — olopatadine hydrochloride ophthalmic solution 0.7%
  Other Names: PAZEO
  Arms: Antihistamine

SUMMARY:
This prospective, open-label, single-center, randomized, investigator-sponsored clinical study seeks to compare patient-reported and clinical outcomes with DEXTENZA versus topical steroid or antihistamine treatment in patients with allergic conjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age
* Provide written informed consent and sign HIPAA form
* Be willing and able to follow all instructions and attend all study visits
* Be able and willing to discontinue wearing contact lenses throughout the study period
* Have a BCVA of ≥50 ETDRS letters (20/100 Snellen equivalent or better) in each eye as measured at Screening visit
* Have urine pregnancy testing for women considered capable of becoming pregnant; not be lactating; and agree to use a medically acceptable form of birth control throughout the study period
* Have a positive history of bilateral ocular allergies and a positive skin test reaction to a perennial allergen and a seasonal allergen as confirmed by the allergy testing at the Screening visit

Exclusion Criteria:

* • Known contraindications or sensitivities to the use of any of the medications required per protocol, including known steroid responders

  * Have any ocular condition that in the opinion of the Investigator could affect the subject's safety or study parameters (including, but not limited to uncontrolled narrow angle glaucoma, severe blepharitis, follicular conjunctivitis, iritis, pterygium, dry eye diagnosis, or active ocular infection)
  * Have a known history of retinal detachment, diabetic retinopathy, or active retinal disease
  * Use of systemic, inhaled, or nasal steroids
  * Use of new systemic antihistamine use within 30 days of Screening visit
  * Use of ocular or topical non-steroidal anti-inflammatory drugs (NSAIDs)
  * Use of lid scrubs
  * Use of decongestants
  * Use of immunotherapeutic agents
  * Use of monoamine oxidase inhibitors (MAOIs)
  * Have a congenital or ocular anomaly or anomaly of the punctum that may preclude placement of DEXTENZA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

PRIMARY OUTCOMES:
Patient-reported treatment preference of self-administered topical therapy versus physician-administered therapy at Day 30 (final visit) | 30 days
  Patient-reported treatment preference of self-administered topical therapy versus physician-administered therapy at Day 30 (final visit)

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center of Florida, Pompano Beach, Florida, United States